CLINICAL TRIAL: NCT05836584
Title: A Randomized Phase II Study of Perioperative Atezolizumab +/- Chemotherapy in Resectable MSI-H/dMMR Gastric and Gastroesophageal Junction (GEJ) Cancer
Brief Title: Testing Immunotherapy (Atezolizumab) With or Without Chemotherapy in Locoregional MSI-H/dMMR Gastric and Gastroesophageal Junction (GEJ) Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-03192; NCI-2023-03192 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA2212 (Other: ECOG-ACRIN Cancer Research Group); EA2212 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2023-04-26; First posted 2023-05-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Clinical Stage I Gastric Cancer AJCC v8; Clinical Stage I Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage II Gastric Cancer AJCC v8; Clinical Stage II Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVA Gastric Cancer AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — atezolizumab; Specimen Handling; Capecitabine; Docetaxel; Fluorouracil; dehydroftorafur; Leucovorin; Lymph Node Excision; Magnetic Resonance Spectroscopy; Oxaliplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (chemotherapy, atezolizumab) (Experimental): NEOADJUVANT THERAPY: Patients receive physician's choice of chemotherapy regimen consisting of FLOT or mFOLFOX or CAPOX in addition to atezolizumab IV on study.
  SURGERY: Patients undergo surgery with lymphadenectomy on study.
  ADJUVANT THERAPY: Patients receive FLOT, mFOLFOX, or CAPOX and atezolizumab IV as in neoadjuvant therapy and then receive atezolizumab IV alone.
  Patients also undergo CT or MRI throughout the trial. Patients may optionally undergo PET/CT and/or collection of blood samples throughout the trial. Patients may also undergo ECHO throughout the trial as clinically indicated.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Drug: Capecitabine; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: Echocardiography Test; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Lymphadenectomy; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Procedure: Positron Emission Tomography; Procedure: Surgical Procedure
- Arm B (atezolizumab) (Experimental): NEOADJUVANT THERAPY: Patients receive atezolizumab IV on study.
  SURGERY: Patients undergo surgery with lymphadenectomy on study.
  ADJUVANT THERAPY: Patients receive atezolizumab IV on study.
  Patients also undergo CT or MRI throughout the trial. Patients may optionally undergo PET/CT and/or collection of blood samples throughout the trial. Patients may also undergo ECHO throughout the trial as clinically indicated.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Lymphadenectomy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Surgical Procedure

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Arm A (chemotherapy, atezolizumab)
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm A (chemotherapy, atezolizumab)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm A (chemotherapy, atezolizumab)
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Arm A (chemotherapy, atezolizumab)
Procedure: Lymphadenectomy — Undergo lymphadenectomy
  Other Names: excision of the lymph node; Lymph Node Dissection; Lymph Node Excision
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
  Arms: Arm A (chemotherapy, atezolizumab)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase II trial compares atezolizumab in combination with chemotherapy (docetaxel, oxaliplatin, leucovorin calcium, fluorouracil, capecitabine) to atezolizumab alone for controlling the growth and/or spreading of the disease in patients with gastric or gastroesophageal junction (JEG) cancer that has not spread from where it first started (local) or only has spread to nearby lymph nodes or tissue (locoregional) and has high microsatellite instability (MSI-H) and mismatch repair deficiency (dMMR). The mismatch repair (MMR) system in the body corrects errors made during the copying of DNA and serves as a proofreading function. If this system isn't working correctly, mutations (changes) in DNA occur which can allow the cancer to grow or spread. This is called dMMR (deficient mismatch repair) . MSI-H describes cancer cells that have a high number of mutations within microsatellites. For example, microsatellite testing that shows mutations in 30% or more microsatellites is called microsatellite instability-high (MSI-H). Microsatellites are short, repeated sequences of DNA. There is evidence that MSI-H/ dMMR gastric or GEJ tumors respond well to immunotherapy. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Docetaxel is in a class of medications called taxanes. It stops tumor cells from growing and dividing and may kill them. Oxaliplatin is in a class of medications called platinum-containing antineoplastic agents. It damages the cell's DNA and may kill tumor cells. Capecitabine is in a class of medications called antimetabolites. It is taken up by tumor cells and breaks down into fluorouracil, a substance that kills tumor cells. Chemotherapy drugs such as leucovorin calcium and fluorouracil work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Using atezolizumab as immunotherapy with and following chemotherapy versus atezolizumab alone prior to and after surgery may shrink or stabilize the tumor in patients with MSI-H/dMMR localized gastric or GEJ cancer and may increase the length of time after treatment that cancer does not come back or get worse.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare three-year event-free survival (EFS) following the administration of perioperative atezolizumab and chemotherapy versus atezolizumab alone in patients with resectable microsatellite instability-high (MSI-H)/mismatch repair deficiency (dMMR) gastric and gastroesophageal junction (GEJ) cancer.

SECONDARY OBJECTIVES:

I. To assess tumor regression grade (TRG) rates following the administration of perioperative atezolizumab and chemotherapy versus atezolizumab in patients with resectable MSI-H/dMMR gastric and gastroesophageal junction (GEJ) cancer.

II. To assess overall survival (OS) following the administration of perioperative atezolizumab and chemotherapy versus atezolizumab in patients with resectable MSI-H/dMMR gastric and gastroesophageal junction (GEJ) cancer.

III. To assess the toxicity associated with the administration of perioperative atezolizumab and chemotherapy versus atezolizumab in patients with resectable MSI-H/dMMR gastric and gastroesophageal junction (GEJ) cancer.

IV. To correlate circulating tumor-derived deoxyribonucleic acid (ctDNA) clearance (defined as > 50% reduction or a reduction to undetectable levels) with TRG, EFS and OS.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A:

NEOADJUVANT THERAPY: Patients receive physician's choice of chemotherapy regimen consisting of 4 cycles of docetaxel intravenously (IV), oxaliplatin IV, leucovorin calcium IV, and fluorouracil IV (FLOT) or 4 cycles of oxaliplatin IV, leucovorin calcium IV, and fluorouracil IV (mFOLFOX) or 3 cycles of oxaliplatin IV and capecitabine orally (PO) (CAPOX) in addition to atezolizumab IV on study.

SURGERY: Patients undergo surgery with lymphadenectomy on study.

ADJUVANT THERAPY: Patients receive FLOT, mFOLFOX, or CAPOX and atezolizumab IV as in Neoadjuvant Therapy and then receive atezolizumab IV alone.

ARM B:

NEOADJUVANT THERAPY: Patients receive 3 cycles of atezolizumab IV on study.

SURGERY: Patients undergo surgery with lymphadenectomy on study.

ADJUVANT THERAPY: Patients receive 9 cycles of atezolizumab IV on study.

All patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial. Patients may optionally undergo positron emission tomography (PET)/CT and/or collection of blood samples throughout the trial. Patients may also undergo echocardiography (ECHO) throughout the trial as clinically indicated.

Patients are followed up for 10 years from the date of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 18 years of age
* Patient must have histologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction adenocarcinoma that is MSI-H/dMMR (microsatellite instability-high/mismatch repair deficient) as determined by one of three methods:

  * Deficient deoxyribonucleic acid (DNA) mismatch repair protein (MMR) expression status: MMR status must be assessed by immunohistochemistry (IHC) for MMR protein expression (MLH1, MSH2, MSH6, PMS2) where loss of one or more proteins indicates dMMR. dMMR may be determined either locally or by site-selected reference lab by Clinical Laboratory Improvement Act (CLIA)-certified assay

    * NOTE: Loss of MLH1 and PMS2 commonly occur together
  * Polymerase chain reaction (PCR) determined microsatellite instability
  * MSI-H tumor status determined by next-generation sequencing
* Patient must have previously untreated localized gastric, or Siewert type II or III GEJ (gastroesophageal junction) adenocarcinoma. Tumors must be staged as T2 or greater primary lesion or be any T stage with the presence of positive locoregional lymph nodes- N+ (clinical nodes) without evidence of metastatic disease

  * Siewert type II tumors: tumors located between 1 cm proximal and 2 cm distal to the GEJ
  * Siewert type III tumors: tumors located between 2 and 5 cm distal to GEJ
* Patient must be amenable to surgical resection with therapeutic intent
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500/mcL (obtained =< 14 days prior to randomization)
* Platelets >= 100,000/mcL (obtained =< 14 days prior to randomization)
* Hemoglobin >= 9 g/dL (obtained =< 14 days prior to randomization)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) OR direct bilirubin =< ULN (for patients with total bilirubin > 1.5 x ULN) (obtained =< 14 days prior to randomization)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]): x =< 3 institutional ULN (obtained =< 14 days prior to randomization)
* Creatinine =< 1.5 x institutional ULN OR glomerular filtration rate (GFR) > 50 mL/min/1.73m^2 (obtained =< 14 days prior to randomization)
* Albumin >= 2.5 g/dL (obtained =< 14 days prior to randomization)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN (unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time [PTT] is within therapeutic range of intended use of anticoagulants) (obtained =< 14 days prior to randomization)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN (unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants) (obtained =< 14 days prior to randomization)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Patient must have no contraindications to receive one of the chemotherapy regimens: FLOT or mFOLFOX / CAPOX
* Patient must not have had prior potentially curative surgery for carcinoma of the stomach/GEJ
* Patient must not receive any other standard anti-cancer therapy or experimental agent concurrently with the study drugs
* Patient must have recovered from clinically significant adverse events of their most recent therapy/intervention prior to randomization
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patient must have chest/abdomen/pelvis CT completed within 4 weeks prior to randomization
* Patient may not have received prior treatment with an immune checkpoint inhibitor (anti-PD-1, anti-PDL-1, anti-PDL-2, anti-CTLA4 monoclonal antibody)
* Patient must not have received any live vaccines within 30 days prior to randomization and while participating in the study. Live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine. Patients are permitted to receive inactivated vaccines and any non-live vaccines including those for the seasonal influenza and coronavirus disease 2019 (COVID-19) (Note: intranasal influenza vaccines, such as Flu-Mist [registered trademark] are live attenuated vaccines and are not allowed). If possible, it is recommended to separate study drug administration from vaccine administration by about a week (primarily, in order to minimize an overlap of adverse events)
* Patient must not have active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain- Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue disease, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis and hepatitis. Patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome are ineligible because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but otherwise are eligible.

  * Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients must not be receiving systemic steroid therapy equivalent to > 10 mg prednisone per day or any other form of immunosuppressive therapy within 7 days prior to randomization. Topical corticosteroid or occasional inhaled corticosteroids are allowed
* Patient must not have known interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity, and must not have a known history of prior pneumonitis requiring treatment with steroids, or any evidence of active, non-infectious pneumonitis
* Patient must not have a known history of active TB (Bacillus Tuberculosis)
* Patient must not have any hypersensitivity to atezolizumab or any of its excipients
* Patient must not have received any prior chemotherapy, targeted small molecule therapy, or radiation therapy for their MSI-H/dMMR gastric and GEJ cancer
* Patient must not have had an allogeneic bone marrow/stem, cell or solid organ transplant
* Patient must not have a history or current evidence of any condition (e.g., known deficiency of the enzyme dihydropyrimidine dehydrogenase [DPD]), therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Patient must not have any condition that would interfere with the cooperation with the requirements of this trial
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse while on protocol treatment. Patients of childbearing potential must continue contraception measures for 5 months after the last dose of atezolizumab and for 9 months after the last dose of chemotherapy. Male patients with partners of childbearing potential must continue contraception measures for 6 months after the last dose of chemotherapy. Patients of childbearing potential must also not breastfeed while on treatment and for 5 months after the last dose of atezolizumab and for 3 months after the last dose of chemotherapy
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* The investigator must declare the chemotherapy regimen their patient will receive (FLOT or mFOLFOX / CAPOX) prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | From randomization to systemic progression of disease that precludes surgery or distant recurrence, or death due to any cause, assessed up to 3 years
  EFS is defined as the time from randomization to an unfavorable event. Hence, occurrences such as local, resectable recurrences, patients' refusal for surgery of resectable tumor, or patients' undergoing definitive therapy such as salvage surgery would not be counted as events for EFS.

SECONDARY OUTCOMES:
Tumor regression grade (TRG) | Up to 10 years
  Will be assessed in the primary tumor using Becker's grading criteria. Fisher's exact test will be used to compare the TRG across the arms.
Overall survival (OS) | From randomization to death from any cause, assessed up to 10 years
  The stratified log rank test will be used to compare OS across the arms.
Incidence of adverse events | Up to 10 years
  All adverse events will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Formal comparison (hypothesis testing) of toxicity rates across the arms is not a primary goal of this trial and the sample size of 240 patients will provide sufficient power for detecting only relatively large differences in adverse events.
Circulating tumor-derived deoxyribonucleic acid (ctDNA) | Up to 10 years
  The proportion of ctDNA clearance on each arm would be correlated with time-to-event (EFS and OS) and binary (TRG) data of the trial. For correlating ctDNA clearance rates and time-to-event data, cox-regression would be used to estimate the correlation magnitude. For correlating ctDNA and binary data, proportions of ctDNA clearances will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Rajdev, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (133):
- United States (133):
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT05836584/ICF_000.pdf